CLINICAL TRIAL: NCT02548832
Title: Effect of Berberine Plus Bezafibrate Administration on the Lipid Profile of Patients With Mixed Dyslipidemia: A Pilot Clinical Trial
Brief Title: Bezafibrate Plus Berberine in Mixed Dyslipidemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Guadalajara (Other)
Responsible Party: Principal Investigator, Esperanza Martínez-Abundis, Dr. Esperanza Martínez-Abundis, University of Guadalajara
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EABYBL
Record Dates: First submitted 2015-09-10; First posted 2015-09-14 (Estimated); Results first posted 2023-02-24 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2022-01

CONDITIONS: Mixed Dyslipidemia
Keywords: Berberine; Bezafibrate
MeSH Terms: interventions — Berberine; Bezafibrate

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Someone of the team make a key number for each patient (36 enrolled, 12 for each intervention), and then put the numbers in to 36 paper envelopes and let the patient chose one. There was double-blind. And the placebo was calcined magnesia.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Berberine (Experimental): Berberine 500 mg with breakfast, meal, and dinner.
  Interventions: Drug: Berberine
- Bezafibrate (Experimental): Bezafibrate 200 mg on breakfast and dinner.
  Interventions: Drug: Bezafibrate
- Berberine plus Bezafibrate (Experimental): Berberine 500 mg with breakfast, meal, and dinner, and bezafibrate 200 mg only on breakfast and dinner.
  Interventions: Drug: Berberine plus Bezafibrate

INTERVENTIONS:
Drug: Berberine — Berberine 1500 mg, each 24 h for 90 days
  1 Berberine capsule 500 mg for breakfast.
  1 Berberine capsule 500 mg for lunch.
  1 Berberine capsule 500 mg for dinner.
  Arms: Berberine
Drug: Bezafibrate — Bezafibrate capsule 400 mg each 24 h for 90 days.
  1 Bezafibrate capsule 200 mg for breakfast.
  1 Bezafibrate capsule 200 mg for dinner.
  Arms: Bezafibrate
Drug: Berberine plus Bezafibrate — Berberine 1500 mg each 24 h for 90 days
  1 Berberine capsule 500 mg for breakfast.
  1 Berberine capsule 500 mg for lunch.
  1 Berberine capsule 500 mg for dinner.
  Bezafibrate 400 mg each 24 h for 90 days.
  1 Bezafibrate capsule 200 mg for breakfast.
  1 Bezafibrate capsule 200 mg for dinner.
  Other Names: Berberine, bezafibrate
  Arms: Berberine plus Bezafibrate

SUMMARY:
Dyslipidemia, is a cardiovascular risk factor of great importance whose prevalence has increased over the last decade. Part of the components of metabolic syndrome and consensus so far contemplated to increased triglycerides (TG) and reduced high-density lipoprotein cholesterol (HDL-C) as part of the elements for classification, which includes mixed dyslipidemia.

Currently, fibrates, such as bezafibrate, are drugs used in treating hypertriglyceridemia, besides reducing the risk of coronary disease. However, although this treatment is safe, it is not without risks; with increased prevalence of adverse effects as the dose thereof is increased or joins combination with a statin drug for the treatment of mixed dyslipidemia long term.

Among the alternative therapies is berberine, which to reduce cholesterol and triglycerides may be useful in combination with bezafibrate in the treatment of mixed dyslipidemia and as an option with lower cost and lower frequency of adverse events.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the effect of berberine plus bezafibrate administration on the lipid profile of patients with mixed dyslipidemia.The investigators will conduct a double-blind randomized pilot clinical trial with parallel groups in men and women aged 30-60 years old with diagnosis of mixed dyslipidemia.

Patients will be assigned to 3 groups:

1. 12 patients will receive berberine, 1500 mg / day
2. 12 Patients will receive bezafibrate 400 mg / day
3. 12 patients will receive a combination of berberine (1500 mg / day) plus bezafibrate (400 mg / day).

All participants will be determined before and after the intervention: lipid profile, total cholesterol (TC), triglycerides (TG), HDL-C, low-density lipoprotein cholesterol (LDL-C), very low-density lipoprotein (VLDL).

Also weight, Body Mass Index (BMI), waist circumference (WC), glucose, systolic blood pressure (SBP), diastolic blood pressure (DBP), creatinine (CR) uric acid (UA) and tolerability.

Statistical analysis was performed upon the sample of subjects.

Previous start the statistical analysis of the groups will proceed to verify the behavior of the distribution of the variables included by Z Kolmogorov-Smirnov goodness of fit.

The distribution of all the variables under this test is cataloged in normal or not normal, which define the type of statistical test would be performed (parametric or non-parametric). However, based on the sample size, non-parametric tests will be those considered most suitable for application.

The data obtained will be expressed and presented using measures of central tendency and dispersion for quantitative (mean and standard deviation) variables and qualitative variables are expressed as frequencies and percentages.

ELIGIBILITY:
Inclusion Criteria:

A. Men and women

B. Accomplished age 30 to 60 years

C. Diagnosis of mixed dyslipidemia established to meet the following criteria:

* Total cholesterol > 5,17 mmol/l.
* Triglycerides > 1,7 mmol/l.

D. BMI of 25 kg / m^2 to 39.9 kg / m^2, weight stable over the past three months, defined as a variability in the lower body weight of 5%.

E. No drug treatment for lipid profile 3 months prior to baseline.

F. Women must ensure a non-hormonal method to avoid pregnancy during the study period.

G. Written information consent

Exclusion Criteria:

A. Removal for informed consent letter

B. Loss of monitoring

C. Presence of serious adverse event

D. Adherence to treatment <80%

E. Consumption of drugs known about lipid profile, glucose metabolism, blood pressure and body weight during the intervention period influence

F. Intolerance or not tolerability or hypersensitivity to the compounds used in the study

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2013-04; Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Esperanza Martínez-Abundis, Principal Investigator — INTEC, CUCS, University of Guadalajara
Locations (1):
- Institute of Experimental and Clinical Therapeutics (INTEC), CUCS, University of Guadalajara, Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 60 subjects were screened. After a selection process and the signature of the consenting letter, 36 patients were included in the study 12 men and 24 women, they were randomized in one of the 3 groups
Groups:
- Berberine: Men and women aged 30 to 60 years with established diagnosis of mixed dyslipidemia:
  Total Cholesterol > 5,17 mmol/L, Triglycerides > 1,7 mmol/L. Berberine 500 mg with breakfast, meal, and dinner, and placebo only on breakfast and dinner
  Berberine Hydrochloride 500 mg oral capsule: Berberine 1500 mg., homologated with placebo each 24 h for 90 days
  1 berberine capsule 500 mg for breakfast and 1 of placebo.
  1 berberine capsule 500 mg for lunch.
  1 berberine capsule 500 mg and 1 placebo for dinner. Homologated with placebo 1 for breakfast and 1 for dinner.
- Bezafibrate: Men and women aged 30 to 60 years with established diagnosis of mixed dyslipidemia:
  Total Cholesterol > 5,17 mmol/L, Triglycerides > 1,7 mmol/L. Placebo 500 mg with breakfast, meal, and dinner, and bezafibrate 200 mg only on breakfast and dinner.
  Bezafibrate 200 mg oral capsule: Bezafibrate capsule 400 mg each 24 h for 90 days.
  1 bezafibrate 200 mg for breakfast.
  1 of bezafibrate 200 mg for dinner.
  Homologated with placebo 1 for breakfast, 1 for lunch and 1 for dinner.
- Berberine Plus Bezafibrate: Men and women aged 30 to 60 years with established diagnosis of mixed dyslipidemia:
  Total Cholesterol > 5,17 mmol/L, Triglycerides > 1,7 mmol/L. Berberine 500 mg with breakfast, meal, and dinner, and bezafibrate 200 mg only on breakfast and dinner.
  Berberine Hydrochloride 500 mg and Bezafibrate 200 mg oral capsules: Berberine hydrochloride capsule 500 and bezafibrate capsule 200 mg each 24 h for 90 days.
  1 berberine and 1 of bezafibrate 200 mg for breakfast
  1 berberine for lunch
  1 berberine and 1 of bezafibrate 200 mg for dinner
Period: Overall Study
Arm/Group | Berberine | Bezafibrate | Berberine Plus Bezafibrate
Started | 12 | 12 | 12
Completed | 10 | 10 | 10
Not Completed | 2 | 2 | 2
Not completed — Lost to Follow-up | 2 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Berberine: Berberine, 1500 mg/day
- Bezafibrate: Bezafibrate, 400 mg/day
- Berberine Plus Bezafibrate: Berberine (1500 mg/day) plus bezafibrate (400 mg/day)
- Total: Total of all reporting groups
Arm/Group | Berberine | Bezafibrate | Berberine Plus Bezafibrate | Total
Number analyzed (Participants) | 12 | 12 | 12 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.4 (8.6) | 44.8 (9) | 46.8 (10.5) | 46 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 10 | 24
  Male | 4 | 6 | 2 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 12 | 12 | 36
  Not Hispanic or Latino | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Mexico | 12 | 12 | 12 | 36
Triglycerides (TG) [Mean (Standard Deviation); unit: mmol/L] | 2.5 (0.8) | 2.2 (0.8) | 2.6 (0.8) | 2.43 (0.8)
Low-density lipoprotein cholesterol (LDL-C) [Mean (Standard Deviation); unit: mmol/L] | 3.7 (0.7) | 3.2 (0.9) | 3.4 (0.6) | 3.43 (0.73)
Total cholesterol (TC) [Mean (Standard Deviation); unit: mmol/L] | 6.0 (0.6) | 6.0 (0.4) | 6.3 (0.7) | 6.1 (0.56)
High-density lipoprotein cholesterol (HDL-C) [Mean (Standard Deviation); unit: mmol/L] | 1.8 (0.4) | 1.6 (0.5) | 1.7 (0.4) | 1.7 (0.43)
Very low density lipoprotein (VLDL) [Mean (Standard Deviation); unit: mmol/L] | 0.5 (0.2) | 0.4 (0.1) | 0.5 (0.2) | 0.46 (0.16)
Glucose [Mean (Standard Deviation); unit: mmol/L] | 5.4 (0.8) | 5.5 (0.5) | 5.5 (0.6) | 5.46 (0.63)
Uric Acid (UA) [Mean (Standard Deviation); unit: mmol/L] | 315.2 (83.3) | 366.5 (59.5) | 303.3 (83.3) | 328.3 (75.3)
Creatinine (Cr) [Mean (Standard Deviation); unit: mmol/L] | 70.7 (26.5) | 70.7 (26.5) | 61.9 (26.5) | 67.76 (26.5)
Body mass index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 30.1 (4.1) | 31.5 (4.3) | 29.0 (3.3) | 30.2 (3.9)
Waist circumference [Mean (Standard Deviation); unit: cm] | 95.6 (9.6) | 99.1 (11.8) | 89.7 (8.4) | 95.1 (9.9)
Body weight [Mean (Standard Deviation); unit: kg] | 77.6 (10.3) | 83.3 (16.3) | 74.6 (6.5) | 78.5 (11.0)
Systolic blood pressure (SBP) [Mean (Standard Deviation); unit: mmHg] | 121 (11) | 124 (11) | 118 (10) | 121 (10.6)
Diastolic blood pressure (DBP) [Mean (Standard Deviation); unit: mmHg] | 76 (6) | 74 (8) | 76 (6) | 75.3 (6.6)

OUTCOME MEASURES:

1. Primary Outcome: Triglycerides After 90 Days
Description: The blood sample for the determination of triglycerides was taken after an overnight fast and was evaluated at baseline and after 90 days by spectrophotometry method.
Time Frame: 90 days
Measure: Mean (Standard Deviation); unit: mmol/L
Groups:
- Bezafibrate: Bezafibrate 200 mg with breakfast and dinner.
Arm/Group | Berberine | Bezafibrate | Berberine Plus Bezafibrate
Number analyzed (Participants) | 10 | 10 | 10
mmol/L | 2.3 (0.9) | 1.1 (0.4) | 1.3 (0.7)

2. Primary Outcome: Total Cholesterol After 90 Days.
Description: The blood sample for the determination of total cholesterol was taken after an overnight fast and was evaluated at baseline and after 90 days by spectrophotometry method.
Time Frame: 90 days
Measure: Mean (Standard Deviation); unit: mM
Arm/Group | Berberine | Bezafibrate | Berberine Plus Bezafibrate
Number analyzed (Participants) | 10 | 10 | 10
mM | 5.3 (0.5) | 5.8 (0.8) | 4.6 (1.2)

3. Primary Outcome: Low Density Lipoprotein Cholesterol (LDL-c) After 90 Days
Description: The blood sample for the determination of low density lipoprotein cholesterol was taken after an overnight fast and was evaluated at baseline and after 90 days by spectrophotometry method.
Time Frame: 90 days
Measure: Mean (Standard Deviation); unit: mM
Arm/Group | Berberine | Bezafibrate | Berberine Plus Bezafibrate
Number analyzed (Participants) | 10 | 10 | 10
mM | 2.8 (0.8) | 2.4 (0.6) | 2.2 (1.3)

4. Primary Outcome: High Density Lipoprotein Cholesterol (HDL-c) After 90 Days
Description: The blood sample for the determination of high density lipoprotein cholesterol was taken after an overnight fast and was evaluated at baseline and after 90 days by spectrophotometry method.
Time Frame: 90 days
Measure: Mean (Standard Deviation); unit: mM
Arm/Group | Berberine | Bezafibrate | Berberine Plus Bezafibrate
Number analyzed (Participants) | 10 | 10 | 10
mM | 1.5 (0.3) | 2.0 (0.3) | 1.8 (0.5)

5. Primary Outcome: Very Low Density Lipoprotein After 90 Days
Description: The blood sample for the determination of VLDL was taken after an overnight fast and was calculated at baseline and after 90 days as triglycerides/5.
Time Frame: 90 days
Measure: Mean (Standard Deviation); unit: mM
Arm/Group | Berberine | Bezafibrate | Berberine Plus Bezafibrate
Number analyzed (Participants) | 10 | 10 | 10
mM | 0.4 (0.1) | 0.2 (0.0) | 0.2 (0.1)

6. Secondary Outcome: Body Weight (BW) After 90 Days
Description: The body weight was evaluated at baseline and after 90 days after an overnight fast, through a bioimpedance digital scale results are reported in kilograms with a decimal.
Time Frame: 90 days
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Berberine | Bezafibrate | Berberine Plus Bezafibrate
Number analyzed (Participants) | 10 | 10 | 10
kg | 75.4 (10.2) | 83.6 (10.7) | 73.0 (6.2)

7. Secondary Outcome: Body Mass Index (BMI) After 90 Days
Description: The BMI was calculated at baseline and after 90 days by the square of the body height, and is universally expressed in units of kg/m^2, resulting from mass in kilograms and height in metres.
Time Frame: 90 days
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Berberine | Bezafibrate | Berberine Plus Bezafibrate
Number analyzed (Participants) | 10 | 10 | 10
kg/m^2 | 29.6 (4.4) | 31.8 (3.4) | 28.4 (2.8)

8. Secondary Outcome: Waist Circumference (WC) After 90 Days
Description: The waist circumference was evaluated at baseline and after 90 days after an overnight fast with a flexible tape in the midpoint between the lowest rib and the iliac crest and is expressed in centimeters.
Time Frame: 90 days
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Berberine | Bezafibrate | Berberine Plus Bezafibrate
Number analyzed (Participants) | 10 | 10 | 10
cm | 94.0 (11.2) | 98.0 (12.0) | 88.7 (9.2)

9. Secondary Outcome: Systolic Blood Pressure After 90 Days
Description: The systolic blood pressure was evaluated at baseline and after 90 days with a digital sphygmomanometer with the subject sited down on a chair after a resting period of 5 minutes on three occasions. The mean of the three measures was considered as the value of SBP. The value was expressed on mmHg.
Time Frame: 90 days
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Berberine | Bezafibrate | Berberine Plus Bezafibrate
Number analyzed (Participants) | 10 | 10 | 10
mmHg | 122 (10) | 122 (13) | 114 (10)

10. Secondary Outcome: Diastolic Blood Pressure After 90 Days
Description: The diastolic blood pressure was evaluated at baseline and after 90 days with a digital sphygmomanometer with the subject sited down on a chair after a resting period of 5 minutes on three occasions. The mean of the three measures was considered as the value of DBP. The value was expressed on mmHg.
Time Frame: 90 days
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Berberine | Bezafibrate | Berberine Plus Bezafibrate
Number analyzed (Participants) | 10 | 10 | 10
mmHg | 73 (8) | 74 (11) | 72 (10)

11. Secondary Outcome: Fasting Serum Glucose (FSG) After 90 Days
Description: The glucose oxidase technique (Beckman Instruments, Inc., Brea, California, USA) was used to determine fasting serum glucose at baseline and after 90 days with an intra- and interassay coefficient of variation of <1.
Time Frame: 90 days
Measure: Mean (Standard Deviation); unit: mM
Arm/Group | Berberine | Bezafibrate | Berberine Plus Bezafibrate
Number analyzed (Participants) | 10 | 10 | 10
mM | 5.6 (0.4) | 5.5 (0.5) | 5.3 (0.3)

12. Secondary Outcome: Uric Acid After 90 Days
Description: The blood sample for the determination of uric acid was taken after an overnight fast and was evaluated at baseline and after 90 days by spectrophotometry method.
Time Frame: 90 days
Measure: Mean (Standard Deviation); unit: mM
Groups:
- Berberine Baseline: Berberine 500 mg with breakfast, meal, and dinner.
Arm/Group | Berberine Baseline | Bezafibrate | Berberine Plus Bezafibrate
Number analyzed (Participants) | 10 | 10 | 10
mM | 285.5 (166.5) | 350.9 (53.5) | 279.5 (89.2)

13. Secondary Outcome: Creatinine After 90 Days
Description: The blood sample for the determination of creatinine was taken after an overnight fast and was evaluated at baseline and after 90 days by spectrophotometry method.
Time Frame: 90 days
Measure: Mean (Standard Deviation); unit: mM
Arm/Group | Berberine | Bezafibrate | Berberine Plus Bezafibrate
Number analyzed (Participants) | 10 | 10 | 10
mM | 53.0 (26.5) | 44.2 (35.4) | 61.9 (35.4)

ADVERSE EVENTS:
Time Frame: adverse events were collected throughout the 90 days of the study
Groups:
- Berberine: 1500 mg berberine each 24 hours
- Bezafibrate: 400 mg bezafibrate each 24 hours
- Berberine Plus Bezafibrate: 1500 mg berberine each 24 hours plus 400 mg bezafibrate each 24 hours
Arm/Group | Berberine | Bezafibrate | Berberine Plus Bezafibrate
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 5/12 | 5/12 | 2/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Berberine (N=12) | Bezafibrate (N=12) | Berberine Plus Bezafibrate (N=12)
Headache (General disorders) | 1 (1) | 2 (2) | 0 (0)
Dyspepsia (General disorders) | 3 (3) | 3 (3) | 2 (2)
Nausea (General disorders) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Time of intervention and the sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2013-09-04): https://cdn.clinicaltrials.gov/large-docs/32/NCT02548832/Prot_SAP_ICF_000.pdf